CLINICAL TRIAL: NCT06467331
Title: The Effect of Hippotherapy on The Development of Life Satisfaction, Health Literacy and Healthism Attitude of Young Adults After Cancer Treatment: Randomized Controlled Experimental Research
Brief Title: The Effect of Hippotherapy on The Development of Life Satisfaction, Health Literacy and Healthism Attitude of Young Adults After Cancer Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Çakmak (Other)
Collaborators: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor-Investigator, Betül Çakmak, RN, PhD, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18.08.2024
Record Dates: First submitted 2024-06-10; First posted 2024-06-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Nursing; Hippotherapy; Life Satisfaction
Keywords: cancer; nursing; life satisfaction; health literacy; Healthism Attitude
MeSH Terms: conditions — Neoplasms; Personal Satisfaction | interventions — Equine-Assisted Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group in which hippotherapy activity will be applied (Experimental): In the implementation of the experimental group, hippotherapy implementation consisting of a total of 5 stations created by the researchers, lasting 30 minutes individually, will be applied to the individuals in the intervention group for 8 weeks, with the participation of the riding coaches. Research data will be collected by the researchers before the implementation (0th), in the 4th and 8th weeks.
  Interventions: Other: Hippotherapy
- The group in which hippotherapy activity will not be applied (No Intervention): In the control group, no interventions will be administered to the participants; data collection will occur solely at the outset (week 0) and at the research period's conclusion (week 8). After completing the main research activities, participants in the control group will be invited to an activity involving horses.

INTERVENTIONS:
Other: Hippotherapy — Hippotherapy, also known as horse-assisted therapy, is a form of animal-assisted therapy. It consists of regularly scheduled sessions designed to enhance functionality in individuals' lives and contribute to their overall health improvement.
  Other Names: activity with horse
  Arms: The group in which hippotherapy activity will be applied

SUMMARY:
This research aims to evaluate the impact of hippotherapy on life satisfaction, health literacy, and health culture among young adults who have undergone cancer treatment. The study underscores the importance of providing support to patients post-cancer treatment. While the literature extensively supports the use of animal-assisted interventions in nursing care plans and practices, there is a notable absence of studies examining the holistic effects of hippotherapy on cancer survivors, both nationally and globally. Given that nurses play a pivotal role in the prevention, diagnosis, treatment, and rehabilitation stages of all diseases, and strive to enhance patient quality of life through comprehensive care, the findings of this project are expected to not only bolster the visibility and professional efficacy of nurses but also inspire similar future research. The research tools employed will determine how complementary supportive practices influence the life satisfaction, health literacy, and health culture of young adults during critical life-shaping periods. These results could provide significant evidence of the nurse's role in patient education, support, and overall care improvement.

DETAILED DESCRIPTION:
Cancer is one of the most important diseases that threaten human health today. It is predicted that the number of cancer survivorship will increase in the future with advances in diagnosis, treatment and care approaches. It is stated that after cancer treatment, individuals have difficulty in continuing treatment due to reasons such as post-treatment side effects, economic and social problems, and their quality of life is negatively affected. It is stated that cancer diagnosis and treatment processes can be observed more specifically in young adults compared to other age groups. It is reported that especially young adults with cancer experience higher levels of depression, worse quality of life and deterioration in body image during treatment, and have difficulty achieving goals related to social, business and academic life. For this reason, it is thought that health professionals have important roles and responsibilities in supporting the lives of young adults, especially after cancer treatment. Nurses should be able to determine the psychosocial needs of individuals, support them in creating positive behavioral changes, empower individuals about coping methods, and take an active role in improving the quality of life of individuals. Complementary methods are one of the approaches frequently included in nurses' care content. Animal-assisted interventions, which are one of the complementary methods, are used at a very limited level in our country. In the Nursing Interventions Classification (NIC) system, it is stated that Animal Assisted Practices contribute positively to the physical, spiritual and social recovery of the individual. Hippotherapy, also known as horse-assisted therapy, is one of the animal-assisted therapies. They are regularly scheduled activities implemented to provide functionality to individuals' lives and contribute to the improvement of their general health status. With these activities, it is aimed to improve the perception of individuals in the sensory field, to strengthen self-confidence, to relax, to provide peace of mind, courage and self-confidence, to remove fear and discouragement, to eliminate distraction, supporting group speaking training, increasing the ability of the individual to express himself, to provide social support for each individual. It aims to ensure that they are always ready for communication. This project will examine the effect of Hippotherapy on life satisfaction, health literacy and the development of a healthy culture of young adult individuals after cancer treatment. The sample of the research will consist of 40 individuals between the ages of 18-35 who have been diagnosed with cancer and completed their treatment. A life satisfaction scale, health literacy scale, health culture scale and qualitative interview form will be used to collect data in the research. In the implementation of the research, hippotherapy implementation consisting of a total of 5 stations created by the researchers, lasting 30 minutes individually, will be applied to the individuals in the intervention group for 8 weeks, with the participation of the riding coaches. Research data will be collected by the researchers before the implementation (0th), in the 4th and 8th weeks of the implementation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30
* He has been diagnosed with cancer and his treatment has been completely completed.
* Least literate
* Pregnant and non-puerperal
* Does not have any physical or cognitive disabilities
* No visual or auditory disabilities

Exclusion Criteria:

* Individuals who cannot participate in all hippotherapy activities

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the health literacy level of young adults with hippotherapy effectiveness | 12 weeks
  The Health Literacy Scale consists of three sub-dimensions: Functional Health Literacy (Items 1, 2, 3, 4, 5), Interactive Health Literacy (Items 6, 7, 8, 9, 10), and Critical Health Literacy (Items 11, 12, 13, 14). Each item on the scale is scored from "strongly disagree" (1 point) to "strongly agree" (5 points) on a five-point Likert scale. Scores on the scale range from 14 to 70. Higher total scores indicate an increase in the level of health literacy. The Cronbach's alpha reliability coefficient of the Health Literacy Scale is 0.85.
Change in the life satisfaction level of young adults with hippotherapy effectiveness | 12 weeks
  The Life Satisfaction Scale consists of a total of 21 items, one of which is reversed. The scale is designed as a five-point Likert type (1=Not at all suitable, 2=Not suitable, 3=Somewhat suitable, 4=Suitable, 5=Completely suitable). Item 6 of the scale is scored in reverse. The possible scores from the Life Satisfaction Scale range from 21 to 105. Higher scores on the scale indicate that the individual has positive perceptions regarding their own life. The scale has five sub-dimensions: the first sub-dimension is general life satisfaction (Items 1, 2, 3, 4, 5, and 6); the second is relationship satisfaction (Items 7, 8, 9, 10, and 11); the third is self-satisfaction (Items 12, 13, 14, and 15); the fourth is social environment satisfaction (Items 16, 17, and 18); and the fifth is job satisfaction (Items 19, 20, and 21). The Cronbach's alpha reliability coefficient of the scale is calculated as .89.
Change in the Healthism Attitude level of young adults with hippotherapy effectiveness | 12 weeks
  The Healthism Attitude scale consists of 14 items, each rated from "completely disagree" (1 point) to "completely agree" (5 points) on a five-point Likert scale. The scale has two sub-dimensions: the Critique of Individual Actions (Items 1, 2, 3, 4, 5, 6, 7, 8) and Judgment sub-dimension (Items 9, 10, 11, 12, 13, 14). As scores on the scale increase, so does the level of knowledge about the culture of being healthy. The internal consistency coefficient of the Healthism Attitude scale is found to be .891.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will not be shared with other researchers.